CLINICAL TRIAL: NCT03400501
Title: Reducing the Risk of Metabolic Decompensation in Adolescents With Poorly Controlled Type 1 Diabetes by Supervised School Administration of Insulin Degludec
Brief Title: Reducing the Risk of Metabolic Decompensation in Diabetic Adolescents by Supervised School Administration of Insulin
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000020909
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin degludec; Insulin Glargine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- subjects receiving insulin degludec (Experimental): Youth aged 8-18 years with T1D whose diabetes is poorly-controlled (A1c ≥8.5%) will receive insulin degludec injections.
  Interventions: Drug: Insulin Degludec
- Subjects receiving insulin glargine (Active Comparator): Youth aged 8-18 years with T1D whose diabetes is poorly-controlled (A1c ≥8.5%) will receive insulin glargine injections.
  Interventions: Drug: Insulin Glargine

INTERVENTIONS:
Drug: Insulin Degludec — Single daily dose of insulin degludec based on their fasting blood glucose levels and current long acting insulin dose
  Other Names: I-degludec
  Arms: subjects receiving insulin degludec
Drug: Insulin Glargine — Single daily dose of insulin glargine based on their fasting blood glucose levels and current long acting insulin dose
  Other Names: I-glar
  Arms: Subjects receiving insulin glargine

SUMMARY:
This is a pilot study to examine and compare the efficacy of supervised injections of long acting insulins degludec and glargine to protect youth with poorly controlled type 1 diabetes (T1D) from development of ketones.

DETAILED DESCRIPTION:
This study will compare the proportion of days with fasting β-hydroxybutyrate levels ≥0.6 mmol/L at the start of the school week following weekend/holiday breaks in subjects who have been randomized to receive daily injections of I-deg or I-glar. Hypothesis: β-hydroxybutyrate levels will be lower in the morning of the first day of the school week in subjects receiving I-deg than in subjects receiving I-glar, since the long half-life of I-deg will compensate for missed insulin doses over the weekend/holidays. To remove variability due to potential non-compliance during the school week, this study will utilize our routine clinical practice of supervised insulin administration and monitoring of blood glucose and ketones during the school day.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of T1D, diagnosed at least 12 months prior to enrollment
* HbA1c ≥8.5%9 and <14% on enrollment
* Taking no medications known to affect blood glucose levels other than insulin.
* Ability to provide participant written informed consent if age 18 years, or parental written informed consent and participant assent if participant is < age 18 before any trial-related activities
* Current regimen includes insulin detemir or I-glar, as long acting insulin
* Willingness to use either I-glar or I-deg pens as basal insulin, and have school personnel supervise administration
* Willingness to have school personnel supervise fasting blood β-hydroxybutyrate levels first thing in the morning at the beginning and end of each school week
* Willingness to have school personnel supervise fasting blood glucose checks daily in the morning on school days, and eat breakfast after the fasting check

Exclusion Criteria:

* Female participants who are pregnant, breast-feeding or planning on becoming pregnant
* Participant (and parent if age <18) unable to read, write, and speak English.
* Adolescents who are home schooled or no longer attending secondary school
* Participant's school is unable to provide personnel to supervise injections of long-acting insulin or measurement blood glucose and β-hydroxybutyrate levels
* Known or suspected allergy to trial medication(s), excipients, or related products.
* Contraindications to study medications, including hypersensitivity to I-deg or one of its excipients, hypersensitivity to I-glar or one of its excipients, and administration of either during episodes of hypoglycaemia

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Lower beta hydroxybutyrate levels | 4 months
  Will test the the hypothesis that β-hydroxybutyrate levels will be lower in the morning (≥0.6 mmol/L) of the first day of the school week in subjects receiving I-deg, since the long half-life of I-deg will compensate for missed insulin doses over the weekend/holidays.

SECONDARY OUTCOMES:
Control of HbA1c levels | 4 months
  Test the hypothesis that the longer duration of action of I-deg will lead to improvements in glycemic control measured by HbA1c (a secondary aim) and fasting glucose.
Measure of beta hydroxybutyrate levels between the 2 groups. | 4 months
  Test the differences in frequency of elevated β-hydroxybutyrate levels when receiving supervised injections of basal insulin versus when not receiving supervised injections between the I-deg and I-glar groups

CONTACTS AND LOCATIONS:
Overall Officials: William Tamborlane, PhD, Principal Investigator — MED School of Medicine
Locations (1):
- Yale University, New Haven, Connecticut, United States